CLINICAL TRIAL: NCT03244098
Title: In-Home Adjustment of New Spinal Cord Injury Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency); The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20009566; 439128 (Other Grant/Funding Number: Craig H Nielson Foundation)
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition Assistance Program (TAP) (Experimental)
  Interventions: Behavioral: Transition Assistance Program
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Transition Assistance Program — TAP caregivers will receive an SCI caregiving guidebook, a 1-hour intervention session by an SCI clinician before hospital discharge, and four 1-hour telehealth clinic-to-home visits at 1, 2, 4, and 6 weeks after discharge by the same clinician
  Arms: Transition Assistance Program (TAP)

SUMMARY:
To improve spinal cord injury (SCI) rehabilitation through stronger informal caregiving, the proposed study will modify and evaluate a telehealth Transition Assistance Program (TAP) for informal caregivers of individuals with SCI during the transition from hospital to home. The TAP was previously developed for stroke caregivers and has been found to decrease caregiver strain and depression. In the proposed study, the TAP will be modified for SCI and implemented at a state-of-the-art SCI rehabilitation facility with a very high volume of SCI treatment and with telehealth technology already in place through which to test the intervention.

DETAILED DESCRIPTION:
SCI Caregivers will be randomly assigned to either the TAP group or to a control receiving the standard care provided by the rehabilitation facility. The TAP begins before discharge and extends across six weeks. It includes three components to improve caregiver mental health and informal care: (1) skill development, (2) education, and (3) supportive problem solving. TAP caregivers will receive an SCI caregiving guidebook, a 1-hour intervention session by an SCI clinician before hospital discharge, and four 1-hour telehealth clinic-to-home visits at 1, 2, 4, and 6 weeks after discharge by the same clinician. Data will be collected from caregivers and individuals with SCI at baseline immediately before discharge and at 2 and 4 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

SCI Patient Inclusion Criteria:

* have a telephone in the home or cellular phone and are able to talk on the phone in English
* are able to provide informed consent
* demonstrate a clinician-rated loss in motor/sensory function on the ASIA scale (i.e., have a spinal cord injury)

Caregiver Inclusion Criteria:

* have a telephone in the home or cellular phone and are able to talk on the phone in English
* are able to provide informed consent
* are a primary caregiver of the individual with SCI
* Caregivers with scores below 10 on the literacy screen will identify a family member or friend to review the guidebook with the caregiver. If no one is identified, the TAP clinician will review the materials with the caregiver and function in that additional capacity

Exclusion Criteria:

* individual with SCI receives his/her primary care from a professional caregiver or other individual outside of the household besides the primary caregiver
* individuals with SCI or caregivers with known current uncontrolled substance dependence, aphasia, anosognosia (deficit in self-awareness), or treatment due to known self-inflicted injury
* individuals living alone
* prisoners
* SCI patient without decision making capacity to consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Zarit Burden Interview - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  22 item self-report measuring perceived burden on a 4 point scale [(1) Never, (2) Sometimes, (3) Quite Frequently, (4) Nearly Always] Given to the caregiver only in all treatment groups.
The Self-Perceived Burden Scale - Patient - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  25 item self-report measuring perceived self-burden on a 5 point scale [(1) None of the time, (2) A little of the time, (3) Some of the time, (4) Most of the time, (5) All of the time] Given to the patient only in all treatment groups.
Short Form - VR 12 Health Survey - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  12 item self-report measuring participant views on his/her own health. Various scales included:
  1. 6 point scale [(1) All of the time, (2) Most of the time, (3) A good bit of the time, (4) Some of the time, (5) A little bit of the time, (6) None of the time]
  2. 5 point scale [(1) Excellent, (2) Very good, (3) Good, (4) Fair, (5) Poor]
  3. 5 point scale [(1) Much Better, (2) Slightly Better, (3) About the Same, (4) Slightly Worse, (5) Much Worse]
  4. 5 point scale [(5) All of the time, (4) Most of the time, (3) Some of the time, (2) A little bit of the time, (1) None of the time]
  5. 3 point scale [(1) Yes, limited a lot, (2) Yes, limited a little, (3) No, Not limited at all]
  Given to both the patient and caregiver in all treatment groups.
SCI-QOL Positive Affect & Well-Being - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  10 item self-report measuring perceived well-being on a 5 point scale [(1) Never, (2) Rarely, (3) Sometimes, (4) Often, (5) Always] Given to both the patient and caregiver in all treatment groups.
Spinal Cord Independence Measure - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  19 item self-report measuring spinal cord injury patient's independence.
  Each item is scored using the following scales [totals range from 0-100]:
  0, 1 0, 1, 2 0, 1, 2, 3 0, 2, 4, 6 0, 5, 8, 10 0, 1, 2, 3, 4 0, 1, 2, 4, 5 0, 2, 4, 6, 8, 10 0, 3, 6, 9, 11, 13, 15 0, 1, 2, 3, 4, 5, 6, 7, 8
  Each item's scale includes descriptive explanations of levels of independence.
  Example:
  0. Requires total assistance
  1. Requires partial assistance; does not clean self
  2. Requires partial assistance; cleans self independently
  4. Uses toilet independently in all tasks but needs adaptive devices or special setting (e.g., bars) 5. Uses toilet independently; does not require adaptive devices or special setting)
  Given to the patient only in all treatment groups.
Revised Scale for Caregiving Self-Efficacy - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  15 item (+4 practice items) self-report measuring perceived self-efficacy on an 11 point scale [from 0 to 100 in increments of 10; ranging from "cannot do at all" (0) to "moderately certain can do" (50) to, "certain can do" (100)] Given to the caregiver only in all treatment groups.
Relationship Assessment Scale - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  7 item self-report measuring perceived relationship between the caregiver and patient on a 5 point scale [ranging from (1) "Not at all" to (5) "Very much"] Given to both the caregiver and patient in all treatment groups.
Exemplary Care Scale - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  11 item self-report measuring perceived quality of care by/from the caregiver on a 4 point scale [(1) Never, (2) Sometimes, (3) Often, (4) Always] Given to both the caregiver and patient in all treatment groups.
Center for Epidemiologic Studies Depression Scale - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  20 item self-report measuring days of depressive symptoms within the last week on a 5 point scale [(0) Not at all or less than 1 day, (1) 1-2 days, (2) 2-4 days, (3) 5-7 days, (4) Nearly every day for 2 weeks] Given to both the caregiver and patient in all treatment groups.
Dissemination & Implementation Questions | One day
  33 item self-report measuring satisfaction with the TAP intervention on a 7 point scale [(1) Never, (2) Rarely, (3) Occasionally, (4) Sometimes, (5) Often, (6) Very Often, (7) Always] as well as three open ended questions.
  Given to the caregiver only in TAP group.
ADAPSS - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  6 item self-report measuring perception of SCI on a 6 point scale [(1) Strongly Disagree, (2) Moderately Disagree, (3) Mildly Disagree, (4) Mildly Agree, (5) Moderately Agree, (6) Strongly Agree]
  Given to only the patient in all treatment groups.
Brief COPE - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  10 item self-report measuring methods of coping on a 4 point scale [(1) I usually don't do this at all, (2) I usually do this a little bit, (3) I usually do this a medium amount, (4) I usually do this a lot]
  Given to both the patient and caregiver in all treatment groups.
Craig Handicap Assessment and Reporting Technique (CHART) Short Form - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  17 item self-report measuring the level of handicap in a community setting including free response of whole numbers (ex: number of times per week left alone), as well as Yes/No/Not Applicable)
  Given to only the patient in all treatment groups.
Cognitive Flexibility Scale - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  12 item self-report measuring cognitive flexibility regarding problem solving on a 6 point scale [(1) Strongly Agree, (2) Agree, (3) Slightly Agree, (4) Slightly Disagree, (5) Disagree, (6) Strongly Disagree]
  Given to both the patient and caregiver in all treatment groups.
Disability Identity and Opportunity Scale - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  23 item self-report measuring attitudes towards being disabled on a 5 point scale [(1) Strongly Disagree, (5) Strongly Disagree]
  Given to only the patient in all treatment groups.
Family Dynamics Scale - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  15 item self-report scale measuring perceived family dynamics (including communication, adaptability, etc.) on a 6 point scale [(1) Extremely Well, (2) Very Well, (3) Well, (4) A Bit, (5) Not Well, (6) Not at All]
  Given only to the caregiver in all treatment groups.
Generalized Anxiety Disorder 7 (GAD 7) - Change from Baseline, at 2 and 4 Months after Discharge | Baseline, 2 months after discharge, 4 months after discharge
  7 item self-report scale measuring level of anxiety over the last 2 weeks on a 4 point scale [(0) Always, (1) Often, (2) Sometimes, (3) Occasionally]
  Given to both the patient and caregiver in all treatment groups.
Spinal Cord Injury Coping Questionnaire - Change from Baseline, at 2 and 4 Months after | Baseline, 2 months after discharge, 4 months after discharge
  12 item self-report scale measuring the acceptance, fighting spirit, and social reliance of an SCI patient on a 4 point scale [(1) Strongly Agree, (2) Agree, (3) Disagree, (4) Strongly Disagree]
  Given to only the patient in all treatment groups
Ten-Item Personality Inventory - Change from Baseline, at 2 and 4 Months after | Baseline, 2 months after discharge, 4 months after discharge
  10 item self-report scale measuring personality (based on the Big 5) on a 7 point scale [(1) Disagree Strongly, (2) Disagree Moderately, (3) Disagree a Little, (4) Neither Agree nor Disagree, (5) Agree a Little, (6) Agree Moderately, (7) Agree Strongly]
  Given to both the patient and caregiver in all treatment groups

SECONDARY OUTCOMES:
Demographics - Patient | Baseline, 2 months after discharge, 4 months after discharge
  34 item self-report demographics survey, including specific information regarding the SCI and relationship between the patient and caregiver.
  16 items on baseline and 18 items for the two follow up sessions.
  Given to the patient only in all treatment groups.
Demographics - Caregiver | Baseline, 2 months after discharge, 4 months after discharge
  31 item self-report demographics survey, including specific information regarding the relationship between the caregiver and patient.
  20 items on baseline and 11 items for the two follow up sessions.
  Given to the caregiver only in all treatment groups.
Brief Health Literacy Screening Tool | One day
  4 item self-report measuring caregiver literacy on a 5 point scale [(1) Always, (2) Often, (3) Sometimes, (4) Occasionally, (5) Never] Given to the caregiver only in all treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Perrin, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perrin PB, McDonald SD, Watson JD, Pierce BS, Elliott TR. Telehealth Transition Assistance Program for Acute Spinal Cord Injury Caregivers: Protocol for a Mixed-Methods, Randomized Controlled Trial. JMIR Res Protoc. 2021 Mar 29;10(3):e28256. doi: 10.2196/28256. PMID 33779569